CLINICAL TRIAL: NCT01022151
Title: Aminophylline Improves Early Postoperative Cognitive Recovery After Sevoflurane Anaesthesia: A Dose-Dependent Study
Brief Title: Aminophylline and Cognitive Function After Sevoflurane Anaesthesia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: King Faisal University (Other)
Responsible Party: Mohamed R. El-Tahan, Department of Anaesthesia and Surgical ICU, Faculty of Medicine, King Faisal University, Dammam, KSA
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 23/2007; 2007 (Other: King Faisal University)
Record Dates: First submitted 2009-11-26; First posted 2009-12-01 (Estimated); Last update posted 2010-11-19 (Estimated); Status verified 2010-11

CONDITIONS: Anaesthesia
Keywords: Aminophylline; sevoflurane; anaesthesia; recovery; cognitive function; entropy
MeSH Terms: interventions — Aminophylline; Doxapram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Placebo [group P] (Placebo Comparator)
  Interventions: Drug: Placebo [group P]
- Aminophylline 2 mg/Kg [group A2] (Active Comparator)
  Interventions: Drug: 0.2 mL/kg of aminophylline 10 mg/mL [group A2]
- Aminophylline 3 mg/Kg [group A3] (Active Comparator)
  Interventions: Drug: 0.2 mL/kg of aminophylline 15 mg/mL [group A3]
- Aminophylline 4mg/Kg [group A4] (Active Comparator)
  Interventions: Drug: 0.2 mL/kg of aminophylline 20 mg/mL [group A4]
- Aminophylline 5 mg/Kg [group A5] (Active Comparator)
  Interventions: Drug: 0.2 mL/kg of aminophylline 25 mg/mL [group A5]
- Doxapram 1 mg/kg [group D] (Active Comparator)
  Interventions: Drug: Doxapram 1 mg/kg [group D]

INTERVENTIONS:
Drug: Placebo [group P] — receive intravenous injection of 0.2 mL/kg of saline 0.9%L [group P]. All study solutions were injected within 1 min at T0 after discontinuation of sevoflurane. No stimulation was applied to patients during this period.
  Arms: Placebo [group P]
Drug: 0.2 mL/kg of aminophylline 10 mg/mL [group A2] — receive intravenous injection of 0.2 mL/kg of aminophylline 10 mg/mL [group A2]. All study solutions were injected within 1 min at T0 after discontinuation of sevoflurane. No stimulation was applied to patients during this period.
  Arms: Aminophylline 2 mg/Kg [group A2]
Drug: 0.2 mL/kg of aminophylline 15 mg/mL [group A3] — receive intravenous injection of 0.2 mL/kg of aminophylline 15 mg/mL [group A3]. All study solutions were injected within 1 min at T0 after discontinuation of sevoflurane. No stimulation was applied to patients during this period.
  Arms: Aminophylline 3 mg/Kg [group A3]
Drug: 0.2 mL/kg of aminophylline 20 mg/mL [group A4] — receive intravenous injection of 0.2 mL/kg of aminophylline 20 mg/mL [group A4]. All study solutions were injected within 1 min at T0 after discontinuation of sevoflurane. No stimulation was applied to patients during this period.
  Arms: Aminophylline 4mg/Kg [group A4]
Drug: 0.2 mL/kg of aminophylline 25 mg/mL [group A5] — receive intravenous injection of 0.2 mL/kg of aminophylline 25 mg/mL [group A5]. All study solutions were injected within 1 min at T0 after discontinuation of sevoflurane. No stimulation was applied to patients during this period.
  Arms: Aminophylline 5 mg/Kg [group A5]
Drug: Doxapram 1 mg/kg [group D] — receive intravenous injection of 0.2 mL/kg of doxapram 5 mg/mL [group D]. All study solutions were injected within 1 min at T0 after discontinuation of sevoflurane. No stimulation was applied to patients during this period.
  Arms: Doxapram 1 mg/kg [group D]

SUMMARY:
Early postoperative recovery of neurologic and cognitive functions is especially advantageous after fast-tracking ambulatory procedures to hasten home discharge after surgery.1 It is well known that volatile anaesthetic agents may generate adverse postoperative cognitive effects and even traces of it may affect task performance in healthy volunteers.2Hence, rapid elimination of the volatile anaesthetics may help reduce postoperative confusion and cognitive impairment in surgical patients by facilitating a faster recovery from general anaesthesia.3 Sevoflurane has been advocated for the routine anesthesia for ambulatory surgery patients. It activates adenosine A1 receptors in primary rat hippocampal cultures through the liberation of adenosine secondary to the interaction of with adenosine transport or key enzymes in adenosine metabolism.4 However; sevoflurane anaesthesia is associated with slower emergence and delayed early postoperative cognitive recovery than desflurane5 and xenon2 anaesthesia.

Aminophylline, which is a hydrophilic cyclic adenosine mono-phosphate (cAMP) dependent phosphodiesterase inhibitor has been used for long time to antagonize the sedative effects of morphine, diazepam, and barbiturates.6-7Aminophylline in doses of 2-5 mg/kg shortens the recovery from sevoflurane anaesthesia and improves bispectral index scores (BIS) with concurrent increases in heart rate which might have a detrimental effect in patients with ischaemic heart disease.8-11However, the use of smaller doses of 2-3 mg/kg is associated with less increases in heart rate. 10-11 The use of 1 mg/kg of Doxapram is comparable to 2 mg/kg of aminophylline in improvement of early recovery from sevoflurane anaesthesia secondary to its central nervous system stimulating effect rather than increased ventilatory elimination of sevoflurane.11 Currently, there is no available published studies have investigated the effects of either theophylline or doxapram on early postoperative cognitive recovery after balanced anaesthesia with sevoflurane.

We hypothesized that the use of small doses of aminophylline [2-3 mg/kg] may be comparable to larger doses in improvement of the early postoperative cognitive recovery from sevoflurane anaesthesia with associated non-significant increases in heart rate.

The present study investigated the effects of 1 mg/kg of doxapram, and 2, 3, 4, and 5 mg/kg of aminophylline on the early postoperative cognitive recovery using the Short Orientation Memory Concentration Test (SOMCT), response entropy (RE) state entropy (SE), difference between RE and SE (RE-SE), end-tidal sevoflurane concentration, haemodynamics, the times to eyes opening and to extubation and degree of sedation after sevoflurane anaesthesia in patients undergoing ambulatory surgery.

DETAILED DESCRIPTION:
One-hundred-eighty ASA I-II patients aged 18-55 years scheduled for elective ambulatory general surgery with a duration >1 h under general anaesthesia were enrolled in this double-blinded placebo-controlled randomised study after obtaining of the approval of Institutional Ethical Committee of author's centre and a written informed consent from the participants.

Based upon our preliminary data, a prior power analysis indicated that 27 patients in each group was a sufficiently large sample size to detect a 20% difference on the Short Orientation Memory Concentration Test (SOMCT)12 at 30 minutes after extubation, with a type-I error of 0.05 and type II error of 0.2. We added 10% more patients to account for patients dropping out during the study. Participants were allocated randomly to six groups (n=30 for each) to receive saline [group P], 1 mg/kg of doxapram [group D] or 2, 3, 4 or 5 mg/kg of aminophylline [groups A2, A3, A4, and A5, respectively] at the end of surgery.

Patients with history of significant cardiovascular, respiratory, cognitive dysfunction, cerebrovascular disease, neurological or psychiatric diseases, pregnancy, and obesity (body mass index ≥ 30 Kg/m2), recent history of infection or recent fever, or adverse reaction to aminophylline or sevoflurane, alcoholism, drug dependence or those receiving xanthines, ß-agonist, anticholinergic, tranquilizers, anticonvulsants or antidepressants or those who has habitual coffee consumption exceeding 2 cups per day, are unable to read, or are suffering from serious hearing or vision impairment were excluded from the study. All operations were performed by the same surgeons.

Primary outcome variable included early postoperative cognitive function. Secondary outcome variables included changes in entropy variables, end-tidal sevoflurane and recovery pattern.

The SOMCT is a patient-based test designed to assess cognitive function in terms of level of orientation, memory, and concentration, The SOMCT requires subjects to recall the current year, and one sentence, and to repeat in numerical order and reverse order the sequence of the months through the year. These six variables yield scores ranging from 0 to 28, with higher scores indicating better function and scores more than 20 were considered normal (Appendix 1).12 A blind investigator who was not involved in the management of the patient and who was blinded to the study drugs explained the SOMCT to the participant and applied it 30 min before induction. All patients received the same explanation of the test by the same investigator.

No premedications were given. A cannula was inserted in a forearm vein and Lactated Ringer's solution was infused at a rate of 2-3 mL/kg/h. Patients monitoring included electrocardiography, pulse oximetry, non-invasive blood pressure and nasopharyngeal temperature monitoring (Datex-OhmedaTM S/5TM, Helsinki, Finland). RE and SE were monitored with the Datex-OhmedaTM S/5 Entropy Module using a specific entropy sensor (M-EntropyTM, Datex-Ohmeda Division, Instrumentarium Corporation, Helsinki, Finland). The sensors were applied appropriately to the patient's forehead according to the manufacturer's instructions. Neuromuscular block were monitored by a train-of-four (TOF) stimulation of the ulnar nerve.

The attending anaesthesiologists who gave the anaesthetic were not involved in the collection of the patient's data. General anaesthesia was induced with propofol (2-3 mg/kg) and fentanyl (2-3 µg/kg). Rocuronium (0.6 mg/kg) was given and tracheal intubation was carried out at the development of maximum block of the TOF. After tracheal intubation, the minimum alveolar concentration (MAC), the end-tidal concentrations of sevoflurane (EtSevo) and end-tidal concentrations of carbon dioxide (EtCO2) were monitored. Anaesthesia was maintained with 0.5-1 MAC of sevoflurane in combination with 50% air in oxygen in a semi-closed circuit with total gas flow of 1 L/min, based on entropy reading where the end-points were SE of ≤ 50 and SE-RE difference less than 10.13 The patient's lungs were ventilated mechanically to maintain the EtCO2 at 35-40 mm Hg. Rocuronium increments were given to maintain suppression of the second twitch using a train-of-four stimulation. Normothermia was maintained using forced-air warming blankets. No supplementary dose of muscle relaxant was administered 30 minutes before the end of the surgery.

During surgery, patients received lornixicam 16 mg and paracetamol 15 mg/kg for postoperative pain relief and granisetron 1 mg for postoperative nausea and vomiting (PONV) prevention.

During skin closure, neuromuscular blockade was antagonized with 50 µg/kg neostigmine and 10 µg/kg glycopyrrolate when the train of four ratio (TOF ratio) ranged between 0.3 and 0.5. At the last skin suture, sevoflurane was discontinued (T0) and the patient's lungs were ventilated with 100% oxygen at 5 litres/min.

Subjects were allocated randomly to six groups (n=30 for each) by drawing sequentially numbered sealed opaque envelopes containing a computer-generated randomisation code to receive intravenous injection of 0.2 mL/kg of a study solution containing either saline 0.9% solution [group P], doxapram 5 mg/mL [group D], or 10 mg/mL [group A2], 15 mg/mL [group A3], 20 mg/mL [group A4], or 25 mg/mL [group A5] of aminophylline. All study solutions were injected within 1 min at T0 after discontinuation of sevoflurane. No stimulation was applied to patients during this period. The test solutions looked identical and contained normal saline, doxapram or aminophylline. They were prepared in identical syringes labelled 'study drug', before induction of anaesthesia by an independent anaesthesiologist who was not involved in the study. The attending anaesthesiologists who were blinded to the study protocol and the patient's randomization code gave the anaesthetic, study solution and established awakening. All staff in the operating room, post anaesthesia care unit (PACU), and day-case surgery ward was unaware of the randomization code.

All measurements were made by the same investigator who was not involved in the management of the patient and who was blinded to the study drugs. Therefore, the patient did not know his/her assigned treatment group. All data, including RE, SE, (RE-SE), the MAC and end-tidal concentration (EtSevo) of sevoflurane, heart rate (HR), and mean arterial blood pressure (MAP) was recorded every 1 min after administration of the study drug (T0) for 15 min.

Tracheal extubation was performed immediately after suctioning when all extubation criteria were achieved (TOF ratio ≥ 0.9, spontaneous ventilation and the ability to follow verbal commands, eye opening, head lift ≥ 5 seconds, and handgrip), at the discretion of the anaesthetist who was involved in the intraoperative management of the patient. The level of consciousness was assessed using simple verbal commands ('open your eyes', 'move your hand') and was repeated up to three times with increasing forcefulness if the subject failed to respond.

Recovery from anaesthesia was assessed by the times to eyes opening (time from T0 to spontaneous eye opening), response time (time from T0 to squeeze the investigator's hand on command), and the time to extubation (time from T0 to tracheal extubation).

After awakening, patients were transferred to the PACU and physical recovery was assessed using the modified Aldrete score14 every 5 minutes after extubation until it reached at least 9 points and the time to reach a score ≥ 9 was recorded. Postoperative analgesia was provided with 0.5 mg/kg intravenous boluses of meperidine as needed to achieve a visual analog pain scale less than 4 points. Heart rate (HR), mean arterial blood pressure (MAP), respiratory rate, peripheral oxygen saturation, and the degree of sedation (four-point verbal rating scores (VRS): awake, drowsy, rousable or deep sleep) were recorded on the patient's arrival and every 15 min until discharge to the ward.

Early postoperative cognitive function was assessed using the SOMCT test, 30 min before induction and 30, 60 and 90 minutes after extubation.

Discharge of patients from the PACU was determined by clinical criteria at the discretion of the attending anaesthetists and no attempt was made to speed up this process. These criteria included alertness and orientation to time and place, conversant and cooperative, stable vital signs for at least 0.5 hour, able to sit up without dizziness and/or nausea, tolerable pain, and a modified Aldrete score ≥ 9. Home readiness was determined by specific clinical criteria, included stable vital signs for at least 1 h, controllable pain by oral analgesics, absent or mild nausea or emesis, ability to walk without dizziness, and ability to retain oral fluids. Actual discharge time was also recorded.15 Times to reach a PACU discharge, home readiness and home discharge and the cost of the study medications were recorded. Postoperative complications included arrhythmia, tremors, vomiting, nausea, seizures, shivering, agitation, or hypoxemia (SpO2<90%) were recorded.

ELIGIBILITY:
Inclusion Criteria:

1. ASA I-II patients
2. aged 18-55 years
3. scheduled for elective ambulatory surgery
4. duration >1 h under general anaesthesia

Exclusion Criteria:

1. cardiovascular diseases
2. respiratory diseases
3. neurological diseases
4. psychiatric diseases
5. pregnancy
6. obesity
7. adverse reaction to aminophylline or sevoflurane
8. receiving xanthines, ß-agonist, anticholinergic
9. history of cognitive dysfunction
10. cerebrovascular disease
11. recent history of infection or recent fever
12. adverse reaction to aminophylline or sevoflurane
13. alcoholism
14. drug dependence
15. those receiving xanthines, ß-agonist, anticholinergic, tranquilizers, anticonvulsants or antidepressants
16. those who has habitual coffee consumption exceeding 2 cups per day
17. unable to read
18. suffering from serious hearing or vision impairment
19. those who had not completed primary school

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2007-11; Primary Completion 2010-07 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
early postoperative cognitive function | 30 min before induction and 30, 60 and 90 minutes after extubation.
  The SOMCT is a patient-based test designed to assess cognitive function in terms of level of orientation, memory, and concentration.

SECONDARY OUTCOMES:
changes in entropy variables, and end-tidal concentration (EtSevo) of sevoflurane, heart rate (HR), and mean arterial blood pressure (MAP) and recovery pattern | 1 min after administration of the study drug (T0) for 15 min.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed R El Tahan, M.D., Principal Investigator — King Faisal University
Locations (1):
- King Faisal University, Khobar, Eastern Province, Saudi Arabia

REFERENCES:
- [Derived] El Tahan MR. Effects of aminophylline on cognitive recovery after sevoflurane anesthesia. J Anesth. 2011 Oct;25(5):648-56. doi: 10.1007/s00540-011-1190-8. Epub 2011 Jul 14. PMID 21755342